CLINICAL TRIAL: NCT06210854
Title: Double-Blind Randomized Phase II Clinical Trial Assessing Jet Administration of pBI-11 for the Treatment of Patients With HPV16/18+
Brief Title: Assessing Jet Administration of pBI-11 for the Treatment of Patients With HPV16/18+
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRMS-83553; IRB00408026 (Other: Johns Hopkins IRB)
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: HPV Infection
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Tropis Experimental (Experimental): Will receive study drug using the Tropis device
  Interventions: Drug: pBI-11
- Stratis Experimental (Experimental): Will receive study drug using the Stratis device
  Interventions: Drug: pBI-11
- Tropis Placebo (Placebo Comparator): Will receive placebo using the Tropis device
  Interventions: Drug: pBI-11
- Stratis Placebo (Placebo Comparator): Will receive placebo using the Stratis device
  Interventions: Drug: pBI-11

INTERVENTIONS:
Drug: pBI-11 — HPV16/18 vaccine
  Other Names: pBI-11 plasmid DNA

SUMMARY:
This is a randomized phase II study. The primary goal of this study is to determine the safety and tolerability of three monthly pBI-11 DNA administrations in each thigh of patients with persistent human papillomavirus 16 (HPV16) and/or human papillomavirus (HPV18+).

DETAILED DESCRIPTION:
This is a randomized phase II study. The primary goal of this study is two-fold; one is to determine the safety and tolerability of three monthly pBI-11 DNA administrations in each thigh of patients with persistent HPV16 and/or HPV18+ < cervical intraepithelial neoplasia 2 (CIN2), wherein either 0.1 mL (0.3 mg) of the plasmid DNA is administered intradermally (I.D.) into each thigh (for a total of 0.6 mg DNA at each visit) using a Pharmajet Tropis device, or 0.5 mL (1.5 mg) of the plasmid DNA is administered intramuscularly (I.M.) into each thigh (for a total of 3 mg DNA at each visit) using a Pharmajet Stratis device; and the other is to evaluate the effect of vaccine on (HPV16/18) viral DNA clearance. Secondary goals are to seek preliminary evidence of prevention of disease progression and assess induction of an HPV16/18-specific immune response to select the appropriate regimen for a subsequent phase III clinical trial. Persistence is defined as positivity on two sequential tests. A total of 72 participants will be enrolled in 4 arms of the study in a 2:1:2:1 ratio (24 patients randomized to the intervention and 12 patient randomized to placebo via Tropis device, and 24 patients randomized to the intervention and 12 patient randomized to placebo via Stratis device).

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have:

   Negative for Intraepithelial Lesions (NEIL), Atypical Squamous Cells of Undetermined Significance (ASC-US), or Low-grade Squamous Intraepithelial Lesion (LSIL) determined by cervical cytology

   AND

   HPV16 and/or 18+ by Roche Cobas 4800, Roche Linear Array HPV Genotyping test, or other FDA-approved HPV genotyping test (Co-infections with HPV types other than HPV16/18 are permissible).
2. Age ≥ 18 years
3. Baseline Eastern Cooperative Oncology Group performance status of 0, 1 at the time of treatment administration.
4. Patients must have adequate organ function at the time of enrollment as defined by the following parameters:

   * White blood cell count ≥ 3,000
   * Absolute lymphocyte number ≥ 500
   * Absolute neutrophil count ≥ 1,500
   * Platelets ≥ 90,000
   * Hemoglobulin ≥ 9
   * Total bilirubin < 3 X the institutional limit of normal
   * Aspartate Aminotransferase (AST)/Alanine Aminotransferase(ALT) < 3 X the institutional limit of normal
   * Creatinine < 2.5 X the institutional limit of normal
5. Women of child-bearing potential must agree to use long acting contraception (e.g. tubal ligation, intrauterine devine or hormonal implant) or two forms of contraception (e.g. barrier method, oral contraceptives) prior to study entry and for 3 months after final vaccination.
6. Ability to understand and the willingness to sign a written informed consent document.
7. Subject is able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

1. Histologic evidence of CIN2, cervical intraepithelial neoplasia 3 (CIN3), adenocarcinoma in situ or malignancy.
2. Patients with a diagnosis of immunosuppression or active systemic use of immunosuppressive medications such as steroids.
3. Patients who are receiving any other investigational agents within 28 days prior to the first dose.
4. Patients with an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
5. Patients with a history of systemic autoimmune disease such as multiple sclerosis or systemic lupus erythematosus (SLE), but exclusive of a history of thyroiditis, psoriasis, Sjrogen's, or inflammatory bowel disease.
6. Patients who are pregnant or breast feeding or plan to become pregnant within five months of first study treatment.
7. Patient with active infection of, or receiving treatment for Human Immunodeficiency Virus (HIV), Hepatitis C Virus (HCV), or Hepatitis B Virus (HBV).
8. History of prior malignancy with disease free interval <5 years; however, individuals with completely resected basal cell or squamous cell carcinoma of the skin within this interval may be enrolled.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 72 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Safety of Vaccination | 12 months
  To determine the safety of repeat administration of pBI-11 DNA vaccine in patients with persistent HPV16/18+ <CIN2. Safety will be determined by tabulating adverse events including vaccine site reactions.
Feasibility of Vaccination | 12 months
  To determine the feasibility of repeat administration of pBI-11 DNA vaccine in patients with persistent HPV16/18+ <CIN2. Feasibility will be estimated as the percentage of participants receiving all three injections of vaccines.
Effect of Vaccination | 6 months
  To assess the effect of pBI-11 vaccination on the clearance of HPV16/18 in cytologic specimens at month 6

SECONDARY OUTCOMES:
Impact of Vaccination on Progression to HPV 16/18 | 12 months
  To assess the impact of vaccination upon progression to HPV16/18 messenger RNA (mRNA)+ CIN2+ by month 12
Levels of HPV16/18 | Baseline, 6 months, and 12 months
  To evaluate the levels and phenotype of circulation HPV16/18 E6/E7-specific T cells in peripheral blood pre- and post-vaccination by each regimen
Changes in Cytopathology | Baseline, 6 months, and 12 months
  To evaluate changes in cytopathology of specimens taken pre- and post-vaccination by each regimen

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Levinson, MD, Principal Investigator — Johns Hopkins University